CLINICAL TRIAL: NCT02386163
Title: Large-scale ex Vivo Expansion and Characterization of Synovial Membrane MSC (SM-MSC) and Infrapatellar Fat Pad MSC (IF-MSC) for Clinical Application
Brief Title: Large-scale ex Vivo Expansion and Characterization of Two Kinds of MSC From Knee for Clinical Application
Status: Completed | Type: Observational
Sponsor: EMO Biomedicine Corporation (Industry)
Collaborators: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EMO-IF-MSC-01
Record Dates: First submitted 2015-03-02; First posted 2015-03-11 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Knee Injuries
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — MSC from synovial membrane and infrapatellar fat pad
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: MSC from synovial membrane and infrapatellar Fat Pad

SUMMARY:
According to many researches, mesenchymal stem cells (MSC) isolated from synovial membrane and infrapatellar fat pad have higher ex vivo proliferation capacity, multipotency and ability to undergo chondrogenesis.

Based on this concept, the investigators plan to get two removed tissues (synovial membrane and infrapatellar fat pad) from patients who have an operation of TKR (Total Knee Replacement). The investigators are going to isolate and expand MSC from these two tissues respectively, and then compare their characterization and potential for clinical application. In the other hand, the investigators plan to build techniques and procedures which comply with "Good Tissue Practices (GTP)".

ELIGIBILITY:
Inclusion Criteria:

Patient who have an total knee replacement surgery

Exclusion Criteria:

Patient who don't sign the agreement

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For patients who have an operation of total knee replacement.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2014-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Compare MSCs from synovial membrane and infrapatellar fat pad | 2 months
  Comparison items include doubling time, phenotype, chondrogenesis and biological activity.

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hung Chang, MD, Ph.D, Principal Investigator — Far Eastern Memorial Hospital; Shing-Mou Lee, Study Chair — EMO Biomedicine Corp.
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan, Taiwan